CLINICAL TRIAL: NCT00012480
Title: Human Sperm Zona Acceptor: Environmental Effects
Brief Title: Effect of Environmental Exposures on the Egg Fertilizing Ability of Human Sperm
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 6100-CP-001
Record Dates: First submitted 2001-03-09; First posted 2001-03-12 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Male Infertility; Testicular Diseases; Urologic and Male Genital Diseases; Lead Poisoning
Keywords: Lead; Male infertility; Gene expression; Economics, Medical
MeSH Terms: conditions — Infertility, Male; Testicular Diseases; Genital Diseases, Male; Lead Poisoning

SUMMARY:
Our data indicate that environmental exposure to the heavy metal lead are more widespread than currently appreciated and that such exposures are associated with the production of human male subfertility. Lead's effects are observed in male partners of infertile couples attending an IVF clinical, in men acting as semen donors in an artificial insemination program and in men representative of the general public. Our goal is to identify the mechanism(s) underlying lead's anti-fertility action.

DETAILED DESCRIPTION:
Our goal is to understand how environmental and occupational exposures to heavy and transition metal ions injure the human male reproductive tract.

The American Urological Association and the American Society for Reproductive Medicine report that ~15% of couples (i.e., more than 6.1 million people in the U.S.) experience infertility at some time. The male is responsible for infertility of 20% of these couples and contributes to the infertility of another 30-40%. However, the cause(s) of male infertility in many cases is unknown. Our data suggest that lead exposures (in the air, in food and in drinking water) underlie a significant fraction of "unexplained" male infertility. We found that blood and seminal plasma lead levels were elevated in 22% of normospermic males from couples seeking infertility treatment, in 29% of semen donors participating in an artificial insemination program and in 23% of unselected semen donors answering an advertisement for research participation. These elevated lead levels were associated with decreased sperm fertility potential in IVF, in artificial insemination and in pregnancy by coitus. The negative effects of lead on sperm function was correlated with expression of specific forms of sperm ion channels (metal binding proteins that allow lead to enter cells), suggesting that such proteins serve as markers for susceptibility or resistance to the reproductive toxic effects of lead. Further, in cases in which human male lead levels changed markedly over time, there were corresponding changes in sperm ion channel, sperm function and sperm fertility potential. These changes were linked to changes in calcium modulated processes in human testis biopsies obtained from infertility patients and could be mimicked in testes of rats experimentally fed lead.

In the current study, we plan to identify changes in gene expression important to the production of the infertile state by comparing the genes expressed in the testis of control and lead exposed rats which are resistant or susceptible to lead. These findings will help to explain how lead exposure kill cells within the testis. We will then determine whether the same changes occur in human testis biopsies and ejaculated sperm from infertile males with high body burdens of lead. The expected outcome of this study is the identification of a possible mechanism explaining male infertility associated with low sperm counts or idiopathic male infertility, tools for diagnosis of male infertility and the hope for rationale treatment.

ELIGIBILITY:
* Otherwise healthy men seeking fertility evaluation, without history of urologic infections or varicocele.
* Non-smokers.
* Occupationally exposed to lead or not exposed to lead.
* Otherwise healthy men undergoing testis biopsy for clinical assessment of spermatogenesis or for sperm retrieval prior to an attempt at assisted reproduction.
* Otherwise healthy men providing semen specimens for clinical analysis prior to an attempt at assisted reproduction.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Benoff, PhD, Principal Investigator — North Shore University Hospital
Locations (3):
- United States (3):
  - University of Southern California Women's and Children's Hospital, Los Angeles, California
  - North Shore University Hospital, Manhasset, New York
  - Copper Hospital and Fertility Testing Laboratory and Sperm Bank, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Benoff S, Cooper GW, Centola GM, Jacob A, Hershlag A, Hurley IR. Metal ions and human sperm mannose receptors. Andrologia. 2000 Sep;32(4-5):317-29. doi: 10.1046/j.1439-0272.2000.00401.x. PMID 11021525
- [Background] Benoff S, Jacob A, Hurley IR. Male infertility and environmental exposure to lead and cadmium. Hum Reprod Update. 2000 Mar-Apr;6(2):107-21. doi: 10.1093/humupd/6.2.107. PMID 10782569
- [Background] Millan C, Sokol RZ, Shi Q, Hurley IR, Centola GM, Ilasi J, Rooney E, Benoff S. Lead induces epigenetic modification of rat testicular gene expression: a DNA microarray study. In: Robaire B, Chemes H, Morales CR, eds. Andrology in the 21st Century. Proceedings of the VII International Congress on Andrology. Short Communications. Englewood, New Jersey: Medimond Publishing Co. Inc. 2001:335-339.
- [Background] Benoff S, Centola GM, Millan C, Napolitano B, Marmar JL, Hurley IR. Increased seminal plasma lead levels adversely affect the fertility potential of sperm in IVF. Hum Reprod. 2003 Feb;18(2):374-83. doi: 10.1093/humrep/deg020. PMID 12571177
- [Background] Benoff S, Cooper GW, Paine T, Hurley IR, Napolitano B, Jacob A, Scholl GM, Hershlag A. Numerical dose-compensated in vitro fertilization inseminations yield high fertilization and pregnancy rates. Fertil Steril. 1999 Jun;71(6):1019-28. doi: 10.1016/s0015-0282(99)00136-3. PMID 10360904